CLINICAL TRIAL: NCT02152098
Title: Skeletal Muscle Strain Injuries and the Connective Tissue: Characterization, Recovery and Optimal Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Collaborators: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Monika Lucia Bayer, PhD, Bispebjerg Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MI-114
Record Dates: First submitted 2014-05-23; First posted 2014-06-02 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Muscle Strain
MeSH Terms: conditions — Sprains and Strains

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Chronic Exercise (Experimental): Chronic Exercise
  Interventions: Procedure: Chronic Exercise
- Acute Early onset of rehabilitation (Experimental): Acute Early onset of rehabilitation
  Interventions: Procedure: Acute Early onset of rehabilitation
- Chronic control (Experimental): Chronic control
  Interventions: Procedure: Chronic Control
- Acute Delayed onset of rehabilitation (Experimental): Acute Delayed onset of rehabilitation
  Interventions: Procedure: Acute Delayed onset of rehabilitation

INTERVENTIONS:
Procedure: Acute Early onset of rehabilitation — Early onset of rehabilitation
  Arms: Acute Early onset of rehabilitation
Procedure: Acute Delayed onset of rehabilitation — Delayed onset of rehabilitation
  Arms: Acute Delayed onset of rehabilitation
Procedure: Chronic Exercise — Exercise
  Arms: Chronic Exercise
Procedure: Chronic Control — Control
  Arms: Chronic control

SUMMARY:
Firstly, the investigators aim to study the biochemical, structural and functional changes associated with acute muscle strain injury in the acute phase and during rehabilitation in vivo. Specific factors present after the injury and their effects on connective tissue cells will be examined in vitro.

Secondly, the investigators will investigate individuals with chronic pain, scar tissue and inferior function after a previous muscle strain injury and test a specific rehabilitation program to alleviate pain and disabilities associated with the preceding muscle injury. The investigators have the following hypotheses:

1. Humoral growth factors and pro-inflammatory macrophages released into the injured area post strain injury stimulate formation of connective tissue in vitro.
2. Early onset of rehabilitation will be superior to a delayed start of rehabilitation for the healing process, in regards to structural improvement of tissue and better clinical function.
3. Scar tissue following a muscle strain injury is characterized by disorganized structure of connective tissue.
4. Mechanical loading in the form of heavy eccentric muscle activity for 12 weeks will lead to a local re-modeling of scar tissue, and result in improved function and reduced symptoms in patients with chronic pain and impaired function after a previous muscle injury.

ELIGIBILITY:
Inclusion Criteria:

* Acute muscle strain injury
* Chronic muscle strain injury
* Age above 18 years

Exclusion Criteria:

* Daily intake of non-steroidal anti-inflammatory drugs (NSAIDs) within three months prior to the injury
* Smoking
* Diabetes
* Connective tissue and/or rheumatic diseases
* Any observed organ dysfunctions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2014-04; Primary Completion 2016-12 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Return to full physical activity | Baseline; Up to 30 weeks (estimated time frame maximum)
  First time the subject is fully fit to take part in all types of physical activity post injury;

SECONDARY OUTCOMES:
Magnetic resonance images | Baseline, 4 weeks, 6 weeks, 12 weeks, 6 months
  Size of injured tissue; Size and location of hematoma; Measurement of muscle perfusion (indication of metabolic activity)
Ultrasound images | Baseline, 7-14 days, 4 weeks, 6 weeks, 12 weeks, 6 months
  Size and location of injury
Ultrasound images | Baseline, 1 week, 2 weeks
  Volume of hematoma
Strength measurements | Baseline, 4 weeks, 6 weeks, 9 weeks, 12 weeks, 6 months
  Strength tests of injured muscle group compared to healthy muscle group on contralateral leg
Structural changes of tissue | Baseline, 12 weeks
  Evaluation of tissue samples from injured muscle before and after rehabilitation program
Aspiration and characterization of inter-/ intramuscular fluid in the injured muscle | Baseline, 3 -14 days
  The aspirated fluid (hematoma/exudate) will be analyzed for released humoral factors, cell types present and its effect on human fibroblast proliferation

OTHER OUTCOMES:
Pain score on the Visual Analog Scale | Baseline, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 weeks
  Each subject is asked to rate his/ her pain level on the Visual Analog Scale during each rehabilitation session at a pre-defined time points during the work-out.
Injury screening questionnaire | Baseline, 1,2,3,4,5,6,7,8,9,10,11,12 weeks, 6 and 12 months
  Each subject is asked to fill out a questionnaire to record the impact of the injury on his/her physical activity and activities of daily living.
Rehabilitation registration | Baseline, 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 weeks
  Each subject is asked to keep a regular training diary of his/ her rehabilitation progress.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sports Medicine Copenhagen, Bispebjerg Hospital, Bispebjerg Bakke 23, Building 8, Copenhagen, Denmark

REFERENCES:
- [Derived] Bayer ML, Hoegberget-Kalisz M, Svensson RB, Hjortshoej MH, Olesen JL, Nybing JD, Boesen M, Magnusson SP, Kjaer M. Chronic Sequelae After Muscle Strain Injuries: Influence of Heavy Resistance Training on Functional and Structural Characteristics in a Randomized Controlled Trial. Am J Sports Med. 2021 Aug;49(10):2783-2794. doi: 10.1177/03635465211026623. Epub 2021 Jul 15. PMID 34264782